CLINICAL TRIAL: NCT01238549
Title: Extending Veteran Participation in the Validation of the SCI-QOL/CAT
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: B7566-R
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries; Quality of Life
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spinal Cord Injury: Participants with SCI

SUMMARY:
The field of spinal cord injury rehabilitation medicine lacks a reliable, patient reported, health-related quality of life measurement tool. The National Institute of Health has provided funding to develop a spinal cord injury-specific, quality of life survey tool in non-Veterans with spinal cord injury called the spinal cord injury-quality of life (SCI-QOL). This quality of life survey asks questions regarding physical/medical, emotional, and social health as it relates to individuals with spinal cord injury.

The purpose of this study is to include a Veteran population in the making of the quality of life survey. Each participant will be asked to complete a packet of quality of life questions. Participants will be given the opportunity to take the survey a second time, either 7-14 days or 5-7 months after the first survey. Taking the survey twice will allow the research team to test the reliability of the survey. Comparing the SCI-QOL with other legacy measures will allow the investigators to test the validity of the survey.

Additionally, the investigators will be testing the SCI-QOL between Veterans and non-Veterans with SCI to determine if there are differences in their self-reported quality of life.

This study will be recruiting participants at the James J. Peters Veterans Affairs Medical Center, Bronx, New York and the James A. Haley Veterans Affairs Hospital, Tampa, Florida.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Veterans with traumatic spinal cord injury
* At least 18 years old
* Persons judged by their primary care doctor to be competent
* Able to read
* Fluent in English.

Exclusion Criteria:

* Veterans with non-traumatic spinal cord injury ("non-traumatic" is defined as any injury from a chronic condition that resulted in decline of function due to the paralysis. These conditions include, but are not limited to: multiple sclerosis, arteriole-venous malformation, nerve impingement syndromes, congenital birth defects, or other)
* Diagnosis of a cognitive impairment (in the clinical chart) such that it limit the subject's ability to read, understand, and respond to statements about quality of life
* Not fluent in English.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans at the James J. Peters Veterans Affairs Medical Center or the James A. Haley Veterans Affairs Hospital with spinal cord injury
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Spungen, EdD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - James A. Haley Veterans' Hospital, Tampa, Florida
  - James J. Peters VA Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from SCI Clinics at the James J. Peters Veterans Affairs Medical Center, Bronx, New York and the James A. Haley Veterans Hospital, Tampa, Florida.
  284 participants signed consent. 248 participants completed the Quality of Life questionnaires.
Period: Overall Study
Arm/Group | Spinal Cord Injury
Started | 284
Completed | 248
Not Completed | 36

BASELINE CHARACTERISTICS:
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 248
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 185
  >=65 years | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.98 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 236
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 218
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 50
  White | 168
  More than one race | 3
  Unknown or Not Reported | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 248

OUTCOME MEASURES:

1. Primary Outcome: SCI-QoL Independence
Description: Average score on a questionnaire about level of independence. The minimum score on the scale is 24.6 and the maximum is 68.9. Fifty is the average score. Values below 50 indicate a worse outcome. Values above 50 represent a better outcome.
Time Frame: Baseline
Population: One participant did not completed item bank or outcomes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 247
units on a scale | 49.9 (10.2)

2. Secondary Outcome: SCI-QoL Ability to Participate in Social Roles and Activities
Description: Average score on a SCI-QoL Ability to Participate in Social Roles and Activities scale. The minimum score on the scale is 25.1 and the maximum is 61.1. A higher score represents better functioning (more ability to participate in social roles and activities).
Time Frame: Baseline
Population: One participant did not completed item bank or outcomes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 247
units on a scale | 45.5 (8.0)

3. Secondary Outcome: SCI-QoL Anxiety
Description: Average score on SCI-QoL Anxiety. The minimum score on the scale is 36.3 and the maximum is 84.2. A higher score represents more anxiety (worse functioning). A lower score represents less anxiety (better functioning).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 248
units on a scale | 48.3 (10.2)

4. Secondary Outcome: SCI-QoL Bowel Management Difficulties
Description: Average score on SCI-QoL Bowel Management Difficulties. The minimum score on the scale is 39.2 and the maximum is 76.3. A higher score represents more bowel management difficulties (worse functioning). A lower score represents fewer bowel management difficulties (better functioning).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 248
units on a scale | 47.5 (9.8)

5. Secondary Outcome: SCI-QoL Bladder Management Difficulties
Description: Average score on SCI-QoL Bladder Management Difficulties. The minimum score on the scale is 39.7 and the maximum is 76.8. A higher score represents more bladder management difficulties (worse functioning). A lower score represents fewer bladder management difficulties (better functioning).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 248
units on a scale | 50.5 (9.6)

6. Secondary Outcome: SCI-QoL Depression
Description: Average score on SCI-QoL Depression. The minimum score on the scale is 38.3 and the maximum is 81.9. A higher score represents more depression (worse functioning). A lower score represents less depression (better functioning).
Time Frame: Baseline
Population: One participant did not completed item bank or outcomes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 247
units on a scale | 47.7 (9.9)

7. Secondary Outcome: SCI-QoL Pain Behavior
Description: Average score on SCI-QoL Pain Behavior. The minimum score on the scale is 38.2 and the maximum is 76.1. A higher score represents more pain behavior (worse functioning). A lower score represents less pain behavior (better functioning).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 248
units on a scale | 53.7 (9.5)

8. Secondary Outcome: SCI-QoL Pain Interference
Description: Average score on SCI-QoL Pain Interference. The minimum score on the scale is 40.2 and the maximum is 79.7. A higher score represents more pain interference (worse functioning). A lower score represents less anxiety (better functioning).
Time Frame: Baseline
Population: One participant did not completed item bank or outcomes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 247
units on a scale | 54.8 (10.2)

9. Secondary Outcome: SCI-QoL Positive Affect and Well-being
Description: Average score on SCI-QoL Positive Affect and Well-being. The minimum score on the scale is 26.7 and the maximum is 68.6. A higher score represents more positive affect and well-being (better functioning).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 248
units on a scale | 55.7 (9.0)

10. Secondary Outcome: SCI-QoL Resilience
Description: Average score on SCI-QoL Resilience. The minimum score on the scale is 16.4 and the maximum is 66.4. A higher score represents more resilience (better functioning).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 248
units on a scale | 53.9 (11.6)

11. Secondary Outcome: SCI-QoL Satisfaction With Social Roles and Activities
Description: Average score on SCI-QoL Satisfaction with Social Roles and Activities. The minimum score on the scale is 28.3 and the maximum is 60.5. A higher score represents more satisfaction with social roles and activities (better functioning).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 248
units on a scale | 47.5 (6.9)

12. Secondary Outcome: SCI-QoL Stigma
Description: Average score on SCI-QoL Stigma. The minimum score on the scale is 37.8 and the maximum is 77.3. A higher score represents more stigma (worse functioning). A lower score represents less stigma (better functioning).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 248
units on a scale | 50.9 (7.9)

13. Secondary Outcome: SCI-QoL Trauma
Description: Average score on SCI-QoL Trauma. The minimum score on the scale is 38.4 and the maximum is 85.2. A higher score represents more trauma (worse functioning). A lower score represents less trauma (better functioning).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 248
units on a scale | 46.8 (10.3)

14. Other Pre Specified Outcome: SCI-QoL Grief Loss
Description: Average score on SCI-QoL Grief Loss. The minimum score on the scale is 30.9 and the maximum is 76.1. A higher score represents more grief/loss (worse functioning). A lower score represents less grief/loss (better functioning).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 248
units on a scale | 46.5 (11.0)

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Spinal Cord Injury
Serious Adverse Events (participants affected / at risk) | 0/248
Other Adverse Events (participants affected / at risk) | 0/248

LIMITATIONS AND CAVEATS:
This study was designed to determine validity and reliability of the SCI QOL in Veterans with SCI. It was not designed to determine their quality of life.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes